CLINICAL TRIAL: NCT02946528
Title: Urgent-start Peritoneal Dialysis to Improve Treatment in ESRD Patients：A Multi-center Clinical Tial
Brief Title: Urgent-start Peritoneal Dialysis in ESRD Patients：A Multi-center Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Ruijin Hospital (Other); Xin Hua Hospital (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Changhai Hospital (Other); Shanghai University of Traditional Chinese Medicine (Other); Shanghai Tong Ren Hospital (Other); Shanghai Jiading District Central Hospital (Other); Shanghai Songjiang District Central Hospital (Unknown); The Affiliated Hospital of Jiangxi University of Traditional Chinese Medicine (Other); Shanghai Punan Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJ20161021USPD
Record Dates: First submitted 2016-10-24; First posted 2016-10-27 (Estimated); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: End-Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Central Venous Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- urgent-start peritoneal dialysis (Experimental): All patients in urgent-start peritoneal dialysis arm initiate peritoneal dialysis as urgent-start dialysis modality.
  Interventions: Device: urgent-start peritoneal dialysis catheter
- urgent-start hemodialysis (Active Comparator): All patients in urgent-start hemodialysis arm initiate hemodialysis as urgent-start dialysis modality.
  Interventions: Device: central venous catheter

INTERVENTIONS:
Device: urgent-start peritoneal dialysis catheter — Patients initiated peritoneal dialysis as urgent-start dialysis modality with a peritoneal dialysis catheter.
  Arms: urgent-start peritoneal dialysis
Device: central venous catheter — Patients initiated hemodialysis as urgent-start dialysis modality with a central venous catheter.
  Arms: urgent-start hemodialysis

SUMMARY:
Within the last decade, urgent-start peritoneal dialysis(PD) has gained considerable interest amongst nephrologists. Several publications have provided assurances that urgent-start PD is indeed feasible and can serve patients well; however, most of the studies have small sample sizes, retrospective design, and the impact of the urgent-start dialysis modality on outcome, especially on short-term complications, has not been directly evaluated. Therefore, we started this multi-centered, prospective, interventional study compared the dialysis-related complications and survival rate directly between urgent-start PD and HD groups with a large sample to determine the feasibility and safety of urgent-start PD as an alternate initial modality of dialysis for patients who require urgent initiation of dialysis therapy.

DETAILED DESCRIPTION:
The prevalence of chronic kidney disease (CKD) and end-stage renal disease (ESRD) is on the rise worldwide. Moreover, many patients who progress to ESRD, even with regular nephrology follow-up, do not have a distinct plan at the time of initiating dialysis therapy, resulting in an urgent need for dialysis. Urgent-start dialysis refers to urgent initiation of dialysis for ESRD patients with no pre-established functional vascular access or peritoneal dialysis (PD) catheter. Hemodialysis (HD) is preferred in most centers with a high rate of central venous catheter (CVC) use at the time of initiating dialysis among HD patients. There is a significantly increased risk of infectious complications, thrombosis, and other complications associated with CVC use which negatively affects patient prognosis. Within the last decade, urgent-start PD has gained considerable interest amongst nephrologists. Several publications have provided assurances that urgent-start PD is indeed feasible and can serve patients well; however, most of the studies have small sample sizes, and the impact of the urgent-start dialysis modality on outcome, especially on short-term complications, has not been directly evaluated. Therefore, we conducted this multicenter, prospective, randomized clinical trial to compare the dialysis-related complications and survival rate directly between urgent-start PD and HD groups with a large sample to determine the feasibility and safety of urgent-start PD as an alternate initial modality of dialysis for patients who require urgent initiation of dialysis therapy.

ELIGIBILITY:
Inclusion criteria

Patients will be eligible to be included in the study only if all of the following criteria are applicable:

1. Age d 18-80 years at the time of signing the informed consent;
2. Diagnosed as ESRD;
3. Requiring urgent initiation of dialysis due to late presentation or rapid progression of renal disease without a pre-established functional dialysis access;
4. Capable of giving signed informed consent.

Exclusion criteria:

Patients will be excluded from the study if any of the following criteria are applicable:

1. patients with severe volume overload with pulmonary edema;
2. patients with severe hyperkalemia (>6.5 mmol/L);
3. patients with uremia encephalopathy;
4. patients with severe liver failure;
5. patients with uncorrectable shock;

(5)patients with severe risk of bleeding or hemorrhagic disease; (6)patients with contraindications of PD including extensive peritoneal fibrosis adhesion, severe skin disease, extensive abdominal infection or extensive abdominal burns, uncorrectable mechanical problems such as herniation of the umbilicus, herniation of the abdomen, bifida of the bladder, valgus of the peritoneum, peritoneal cavity and chest leakage; (7)patients with Intracranial hemorrhage or increased intracranial pressure; (8)patients with uncorrectable shock; (9)patients who cannot establish a vascular access; (10)patients with malignancy; (11)patients with mental disorder; (12)patients with pregnancy or lactation; (13)patients unable or unwilling to provide informed consent for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
the incidence of dialysis-related complications | 12 months
  the incidence of dialysis-related complications.Dialysis-related complications were defined as a composite of non-infectious complications (malposition, obstruction, leakage, hernia, bleeding, or thrombosis) and infectious complications (catheterrelated infection, exit-site infection, or peritonitis)

SECONDARY OUTCOMES:
PD catheter technical survival rate | 12 months
  PD catheter technical survival rate
peritonitis-free survival rates | 12 months
  peritonitis-free survival rates
patient survival rate | 12 months
  patient survival rate
total medical cost of initial hospitalization | 6 weeks
  total medical cost of initial hospitalization
duration of initial hospitalization | 6 weeks
  duration of initial hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Ni, Doctor, Study Chair — Renji Hospital, School of Medicine, Shanghai Jiao Tong University; Gengru Jiang, Doctor, Principal Investigator — Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine; Niansong Wang, Doctor, Principal Investigator — The Sixth People's Hospital Affiliated to Shanghai Jiao Tong University; Zhiyong Guo, Doctor, Principal Investigator — Changhai Hospital; Xiaonong Chen, Doctor, Principal Investigator — Ruijin Hospital; Feng Ding, Doctor, Principal Investigator — No.9 People Hospital Affiliated to Shanghai Jiao Tong University School of Medicine; Weijie Yuan, Doctor, Principal Investigator — Shanghai General Hospital affiliated to Shanghai Jiao Tong University; Yueyi Deng, Doctor, Principal Investigator — Long Hua Hospital Shanghai University of Traditional Chinese Medicine; Xiaoxia Wang, Principal Investigator — Tong Ren hospital Shanghai Jiao Tong university school of medicine; Ying Li, Principal Investigator — Jiading district central hospital of Shanghai; Xiujuan Zang, Principal Investigator — hanghai Songjiang District Central Hospital; Guoqing Wu, Principal Investigator — The Affiliated Hospital of Jiangxi University of Traditional Chinese Medicine
Locations (1):
- RenJi Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghaffari A. Urgent-start peritoneal dialysis: a quality improvement report. Am J Kidney Dis. 2012 Mar;59(3):400-8. doi: 10.1053/j.ajkd.2011.08.034. Epub 2011 Oct 22. PMID 22019332
- [Background] Alkatheeri AM, Blake PG, Gray D, Jain AK. Success of Urgent-Start Peritoneal Dialysis in a Large Canadian Renal Program. Perit Dial Int. 2016 Mar-Apr;36(2):171-6. doi: 10.3747/pdi.2014.00148. Epub 2015 Sep 15. PMID 26374834
- [Background] Wong LP, Li NC, Kansal S, Lacson E Jr, Maddux F, Kessler J, Curd S, Lester K, Herman M, Pulliam J. Urgent Peritoneal Dialysis Starts for ESRD: Initial Multicenter Experiences in the United States. Am J Kidney Dis. 2016 Sep;68(3):500-2. doi: 10.1053/j.ajkd.2016.03.426. Epub 2016 May 11. No abstract available. PMID 27178678
- [Background] Povlsen JV, Ivarsen P. How to start the late referred ESRD patient urgently on chronic APD. Nephrol Dial Transplant. 2006 Jul;21 Suppl 2:ii56-9. doi: 10.1093/ndt/gfl192. PMID 16825263
- [Background] Ivarsen P, Povlsen JV. Can peritoneal dialysis be applied for unplanned initiation of chronic dialysis? Nephrol Dial Transplant. 2014 Dec;29(12):2201-6. doi: 10.1093/ndt/gft487. Epub 2013 Dec 17. PMID 24353321
- [Background] Koch M, Kohnle M, Trapp R, Haastert B, Rump LC, Aker S. Comparable outcome of acute unplanned peritoneal dialysis and haemodialysis. Nephrol Dial Transplant. 2012 Jan;27(1):375-80. doi: 10.1093/ndt/gfr262. Epub 2011 May 28. PMID 21622993
- [Background] Lobbedez T, Lecouf A, Ficheux M, Henri P, Hurault de Ligny B, Ryckelynck JP. Is rapid initiation of peritoneal dialysis feasible in unplanned dialysis patients? A single-centre experience. Nephrol Dial Transplant. 2008 Oct;23(10):3290-4. doi: 10.1093/ndt/gfn213. Epub 2008 Apr 19. PMID 18424817
- [Background] Povlsen JV, Sorensen AB, Ivarsen P. Unplanned Start on Peritoneal Dialysis Right after PD Catheter Implantation for Older People with End-Stage Renal Disease. Perit Dial Int. 2015 Nov;35(6):622-4. doi: 10.3747/pdi.2014.00347. PMID 26702001
- [Background] Liu Y, Zhang L, Lin A, Ni Z, Qian J, Fang W. Impact of break-in period on the short-term outcomes of patients started on peritoneal dialysis. Perit Dial Int. 2014 Jan-Feb;34(1):49-56. doi: 10.3747/pdi.2012.00293. PMID 24525597
- [Background] Arramreddy R, Zheng S, Saxena AB, Liebman SE, Wong L. Urgent-start peritoneal dialysis: a chance for a new beginning. Am J Kidney Dis. 2014 Mar;63(3):390-5. doi: 10.1053/j.ajkd.2013.09.018. Epub 2013 Nov 15. PMID 24246221
- [Derived] Htay H, Johnson DW, Craig JC, Teixeira-Pinto A, Hawley CM, Cho Y. Urgent-start peritoneal dialysis versus haemodialysis for people with chronic kidney disease. Cochrane Database Syst Rev. 2021 Jan 27;1(1):CD012899. doi: 10.1002/14651858.CD012899.pub2. PMID 33501650
- [Derived] Htay H, Johnson DW, Craig JC, Teixeira-Pinto A, Hawley CM, Cho Y. Urgent-start peritoneal dialysis versus conventional-start peritoneal dialysis for people with chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 15;12(12):CD012913. doi: 10.1002/14651858.CD012913.pub2. PMID 33320346